CLINICAL TRIAL: NCT05437614
Title: Comparison of Outcome and Effectiveness Between Micropulse Diode Laser Cyclophotocoagulation and Cyclocryoablation in Treatment of Refractory Glaucoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Mariam Noor, Post Graduate Trainee, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniversityHSL786
Record Dates: First submitted 2022-06-05; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Treatment of Refractory Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment of refractory glaucoma using Micropulse diode laser cyclophotocoagulation (Active Comparator)
  Interventions: Procedure: Micropulse diode laser cyclophotocoagulation in treatment of refractory Glaucoma
- Treatment of refractory glaucoma using cyclocryoablation (Active Comparator)
  Interventions: Procedure: Cyclocryoablation in treatment of refractory Glaucoma

INTERVENTIONS:
Procedure: Micropulse diode laser cyclophotocoagulation in treatment of refractory Glaucoma — Treatment of refractory Glaucoma by Micropulse diode laser cyclophotocoagulation
  Arms: Treatment of refractory glaucoma using Micropulse diode laser cyclophotocoagulation
Procedure: Cyclocryoablation in treatment of refractory Glaucoma — Treatment of refractory Glaucoma by cyclocryoablation
  Arms: Treatment of refractory glaucoma using cyclocryoablation

SUMMARY:
laucoma having bad prognosis after maximally tolerated medication,glaucoma that fails after filtering operations, neovascular glaucoma, glaucoma following vitrectomy and glaucoma secondary to uveitis etc. is collectively termed as refractory glaucoma. For such glaucoma patients, cyclodestructive procedures are often used to reduce IOP, as well as to relieve ocular and periocular pain. Recently,diode laser transscleral cyclophotocoagulation has proved to be an effective method for the treatment of refractory glaucoma and it has become a standard treatment for refractory glaucoma.(Yu, Q., Liang, Y., Ji, F. and Yuan, Z.,et al 2020. ) In previous articles, little is known about the long-term outcomes of micropulse diode laser cyclophotocoagulation and cyclocryotherapy. Discrepancies in the results of several large observational analyses have introduced further ambiguity on the role of micropulse diode laser cyclophotocoagulation and cyclocryotherapy.The mechanism of transcleral cyclophotocoagulation IOP lowering in refractory glaucoma is not well understood. In this study, we perform cyclocryoablation and micropulse diode laser cyclophotocoagulation in patients with refractory glaucoma and report the outcomes / mechanism of IOP control using this new surgical paradigm. The objective of our project is to assess the end result and outcome of the role of micropulse diode laser cyclophotocoagulation and cyclocryotherapy.We aim to evaluate the comparison between micropulse diode laser cyclophotocoagulation and cyclocryotherapy.

Only those subjects will be recruited who provide written informed consent. Patients are diagnosed on bases of tonometry, gonioscopy, ophthalmoscopy, perimetry. Patients' age, gender, type of glaucoma, number of diode laser treatment sessions, postoperative complications, number of hypotensive medications required to control IOP, and best corrected visual acuity (BCVA) will be evaluated. The criteria for success will be defined as postoperative IOP <21 mmHg or >20% decrease in IOP with or without additional medical treatment.

ELIGIBILITY:
Inclusion Criteria:

Positive diagnosis of refractory glaucoma

* Poor visual acuity: Hand movements or less
* Age ≥ 18 years
* Intraocular pressure ≥ 21 mmHg
* Signed informed consent

Exclusion Criteria:

* Eye surgery performed over the last 3 months
* Eye inflammation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
postoperative complications | 1 year
  Hypotony, Fibrinous uveitis, Cystoid macular edema
Reduced IOP | 1 year
  Reduction in IOP to less than 21 mmHg medications required to control IOP
Decrease in number of hypotensive drugs | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Holy Family Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided